CLINICAL TRIAL: NCT01113684
Title: Clinical and Neurophysiological Study of Subthalamic Brain Stimulation in PD
Brief Title: Study of Subthalamic Brain Stimulation in Parkinson Disease (PD)
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Harrison Walker, MD, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F091215017; 1K23NS067053-01 (NIH)
Record Dates: First submitted 2010-04-26; First posted 2010-04-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Implantable pulse generator (deep brain stimulator) — This study evaluates the effects of subthalamic deep brain stimulation on central and peripheral nervous system activity in patients who have already had brain stimulators placed as a matter of routine clinical care.
  Other Names: Soletra Implantable Pulse Generator (Medtronic, Inc.); Kinetra Implantable Pulse Generator (Medtronic, Inc.); Activa PC Implantable Pulse Generator (Medtronic, Inc.); Activa RC Implantable Pulse Generator (Medtronic, Inc.)

SUMMARY:
Deep brain stimulation (DBS) improves debilitating symptoms of movement disorders when conventional medical therapies and novel surgical therapies fail. Despite the remarkable efficacy of DBS, its therapeutic mechanism remains unclear. There is controversy regarding whether the therapeutic effects of DBS are associated with inhibition or excitation of target neurons, the introduction of new activity into the network, or a combination of these mechanisms. Additionally, it is unclear why stimulus frequency plays an important role in the clinical response to therapy. The fundamental hypothesis of this proposal is that unilateral subthalamic nucleus (STN) DBS in PD alters neuronal activity in the bilateral basal ganglia-thalamic-cortical motor system in a manner that is dependent on stimulation frequency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson disease who have undergone subthalamic deep brain stimulation

Exclusion Criteria:

* Patients who are unable to follow verbal instructions
* Patients who are unable to tolerate being off their Parkinson's medications for 12 hours
* Patients who are medically unstable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease who have undergone subthalamic deep brain stimulation
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
This study measures neurophysiological responses to subthalamic deep brain stimulation in the central and peripheral nervous system in patients with Parkinson disease. | Population data will be analyzed for the primary endpoint in 12 months and reported in approximately 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison C Walker, MD, Principal Investigator — University of Alabama at Birmingham, Department of Neurology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Walker HC, Watts RL, Guthrie S, Wang D, Guthrie BL. Bilateral effects of unilateral subthalamic deep brain stimulation on Parkinson's disease at 1 year. Neurosurgery. 2009 Aug;65(2):302-9; discussion 309-10. doi: 10.1227/01.NEU.0000349764.34211.74. PMID 19625909